CLINICAL TRIAL: NCT01515839
Title: Brain Single Photon Emission Computed Tomography and Quantitative Electroencephalography In Former NFL Players: A Single-Site Exploratory Pilot Study
Brief Title: Single Photon Emission Computed Tomography (SPECT) Imaging Study of Professional American Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amen Clinics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISCAN 001
Record Dates: First submitted 2010-10-01; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Traumatic Brain Injury
Keywords: SPECT; Imaging; Football; Traumatic brain injury; Regional cerebral blood flow
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Fatty Acids, Omega-3; Acetylcarnitine; Ginkgo biloba extract; Thioctic Acid; huperzine A; Acetylcysteine; Phosphatidylserines; vinpocetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supplement intervention (Experimental): Dietary Supplement: Multivitamin, Omega 3 Supplement, Brain and Memory Formula
  Interventions: Dietary Supplement: Multivitamin Supplement intervention

INTERVENTIONS:
Dietary Supplement: Multivitamin Supplement intervention — We recommend the following protocol:
  1. 2 tablets of a high quality multivitamin BID
  2. 2 capsules of omega 3 fish oil BID for a total of 3 grams daily
  3. 3 capsules of a brain and memory formula BID which contains Acetyl-L-Carnitine (HCL) 1000 mg, Ginkgo Biloba Extract 120 mg, Alpha-Lipoic Acid (ALA) 300 mg, Huperzine A (Huperzia serrata)150 mcg, N-Acetyl-L-Cysteine (NAC) 600mg, Phosphatidyl Serine (soy) 100 mg, Vinpocetine 15mg
  4. Weight loss
  Other Names: Omega 3 Fatty Acid; Acetyl-L-Carnitine (HCL); Ginkgo Biloba Extract; Alpha-Lipoic Acid (ALA); Huperzine A (Huperzia serrata); N-Acetyl-L-Cysteine; Phosphatidyl Serine; Vinpocetine

SUMMARY:
The investigators primary objective is to acquire preliminary data on one-hundred former NFL veterans with at least one full year of professional service using brain SPECT imaging in order to assess the degree to which NFL football puts players at risk for traumatic brain injury (TBI). TBI severity shall be gauged via visual inspection by a clinician trained in neuroanatomy, and also by a statistical comparison of subjects' brains to an in-house proprietary database comprised of the brains of healthy subjects.

The investigators secondary objective is to acquire additional data on these players such that investigators may establish causative factors and risks associated with said TBI.

The investigators tertiary objective is to acquire data on subjects using various mental health metrics in order to determine the effects of TBI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Each subject must have been on an active NFL roster for a minimum of one year

Exclusion Criteria:

* Any subjects who could not cease taking psychoactive medications (recreational or otherwise) for an appropriate washout period prior to scanning were excluded from the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
A concentration SPECT scan will be given to assess the changes in regional cerebral blood flow to the brain in our study participants. | The SPECT scan is one day imaging exam. A follow up scan will be performed following a 2-12 month supplement intervention.
  For the concentration study the subject will start the Conner's Continuous Performance Task, a 15-minute computer-administered test of attention, subsequent to the accommodation period. Three minutes into task performance 20 milliCuries of Tc-99m-hexamethylpropylene amine oxime will be injected through the catheter with attention to minimal disruption of the subject's attention task. The subject will proceed to completion of the attention task. The concentration scans will then be compared to a healthy brain subject normative database.

SECONDARY OUTCOMES:
Quantitative electroencephalography (QEEG) will be used to assess the damage to neural networks in our study participants. | The QEEG testing is one day exam. A follow up test will be performed following a 2-12 month supplement intervention.
  Subjects will undergo quantitative electroencephalography (QEEG) testing in both the eyes open and eyes closed condition to measure the electrical activity patterns of the brain. Brain maps will be generated and compared against a normative database.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Amen, MD, Principal Investigator — Amen Clinics, Inc.
Locations (1):
- Amen Clinics, Inc., Newport Beach, California, United States

REFERENCES:
- [Result] Amen DG, Newberg A, Thatcher R, Jin Y, Wu J, Keator D, Willeumier K. Impact of playing American professional football on long-term brain function. J Neuropsychiatry Clin Neurosci. 2011 Winter;23(1):98-106. doi: 10.1176/jnp.23.1.jnp98. PMID 21304145
- [Result] Amen DG, Wu JC, Taylor D, Willeumier K. Reversing brain damage in former NFL players: implications for traumatic brain injury and substance abuse rehabilitation. J Psychoactive Drugs. 2011 Jan-Mar;43(1):1-5. doi: 10.1080/02791072.2011.566489. PMID 21615001